CLINICAL TRIAL: NCT01358357
Title: A Randomized, Double-blind, Placebo-controlled, Flexible-dose, Parallel-group Study of Lurasidone Adjunctive to Lithium or Divalproex for the Prevention of Recurrence in Subjects With Bipolar I Disorder
Brief Title: Bipolar Maintenance Study of Lurasidone Adjunctive to Lithium or Divalproex
Acronym: PERSIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1050296; 2011-000986-10 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Results first posted 2016-07-26 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Bipolar I Disorder
Keywords: Lurasidone; Latuda; Bipolar I
MeSH Terms: interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lurasidone 20-80 mg flexible dose (Experimental)
  Interventions: Drug: Lurasidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 20 mg daily (days 1-3), Lurasidone 40 mg daily (days 4-7), Lurasidone 20-80 mg daily (flexible dose) thereafter
  Arms: Lurasidone 20-80 mg flexible dose
Drug: Placebo — 20-80 mg flexible dose
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, placebo-controlled, flexible-dose, parallel-group study designed to evaluate the efficacy and safety of lurasidone (in combination with lithium or divalproex) for the maintenance treatment of bipolar I disorder in subjects with or without rapid cycling and /or psychotic features.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy and safety of lurasidone (in combination with lithium or divalproex) for the maintenance treatment of bipolar I disorder in subjects with or without rapid cycling and/or psychotic features.

ELIGIBILITY:
Inclusion Criteria:

Open-label Phase

* 18 years of age or older
* Diagnostic and Statistical Manual of Mental Disorders, 4th Ed., Text Revision (DSM-IV-TR) diagnosis of bipolar I disorder

  •≥ 1 manic, mixed manic, or depressed episode in past 2 years
* YMRS or MADRS total score ≥ 14 if on lithium or divalproex; ≥ 18 if not on lithium or divalproex

Double-blind Phase

Inclusion Criteria:

* Subjects must achieve consistent clinical stability, defined as total scores ≤ 12 on the YMRS and MADRS over at least 12 weeks, with the allowance of two excursions (YMRS and/or MADRS total scores up to 13 or 14, respectively) except during the last 4 weeks before randomization

Exclusion Criteria:

Open Label Phase

* Diagnosis of an Axis I or Axis II disorder, other than bipolar I disorder, that is the primary focus of treatment within 3 months of screening
* Subjects for whom diagnostic agreement between the Investigator and United BioSource Corporation (Boston) (UBC) cannot be reached
* Ultra-fast rapid cycling (defined as ≥ 8 mood episodes over the previous 12-month period)
* Subjects who test positive for drugs of abuse at screening. In the event a subject tests positive for cannabinoids (tetrahydrocannabinol), the Investigator will evaluate the subject's ability to abstain from cannabis during the study
* Unstable/inadequately treated medical illness
* The subjects answers "yes" to "Suicidal Ideation" items 4 or 5 on the C-SSRS (at time of evaluation)

Double Blind Phase

* Subjects who in the Investigator's judgment have not been compliant with study medication during the stabilization phase
* Subjects who have not stabilized during the open-label phase (within 20 weeks)
* Subjects who test positive for drugs of abuse at double-blind phase baseline. In the event a subject tests positive for cannabinoids (tetrahydrocannabinol), the Investigator will evaluate the subject's ability to abstain from cannabis during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 965 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (105):
- United States (26):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Behavioral Research Specialists, LLC, Glendale, California
  - AXIS Clinical Trials, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - Stanford University School of Medicine Research Program VA Palo Alto Health Care System, Palo Alto, California
  - SF-CARE, Inc., San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - "Stanford University School of Medicine, Stanford, California
  - Florida Clinical Research LLC, Bradenton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Galiz Research, Miami Springs, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Clinco, Terre Haute, Indiana
  - ActivMed Practices & Research Inc., Haverhill, Massachusetts
  - Psych Care Consultants Research, St Louis, Missouri
  - Village Clinical Research Inc,, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Charak Center for Health and Wellness, Garfield Heights, Ohio
  - Cutting Edge Research Groupd, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Psychoneuroendocrinology Research Group, Dept of Psychiatry, UT Southwestern Medical Center, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
- Argentina (8):
  - Sanatorio Morra, Córdoba, Córdoba Province
  - Centro de Atencion E Invest. Clinica (CAICI), Rosario, Santa Fe Province
  - Novain Neurociencias Group, Buenos Aires
  - Centro de Neuropsiquiatria, Buenos Aires
  - IPEM-Instituto de Prevención de las Enfermedades Mentales., Buenos Aires
  - Instituto DAMCI, Córdoba
  - Clinica Privada de Salud Mental Santa Teresa de Avila, La Plata
  - Centro de Psiquiatria Biologica, Mendoza
- Australia (4):
  - The Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - RWF Medic Pty Ltd as Trustee for Farnbach Family Trust at Neurotherapy Victoria, Malvern, Victoria
  - The Melbourne Clinic, Richmond, Victoria
  - Hollywood Medical Centre, Fremantle, Western Australia
- Bulgaria (6):
  - Psychiatry Dispensary, Burgas
  - University Multiprofiled Hospital for Active Treatment "Sveti Georgi", Plovdiv
  - Regional Psychiatric Dispensary, Rousse
  - Multiprofiled Hospital for Active Treatment "Alexandrovska", Sofia
  - Psychiatric Clinic, Military Medical Academy, Sofia
  - Multprofiled Hospital for Active Treatment "Sveta Marina", Varna
- Chile (3):
  - CETEP, Santiago
  - Clinica Las Condes, Santiago
  - Psicomedica, Santiago
- Croatia (5):
  - Clinic Hospital Centre Rijeka Clinic for Psychiatry, Rijeka
  - Clinical Hospital Centre Zagreb, Zagreb
  - Klinicki Bolnicki Centar Zagreb-Rebro, Zagreb
  - University Hospital Sestremilosrdnice, Zagreb
  - University Hospital Centre Zagreb, Zagreg
- Czechia (11):
  - Saint Anne s.r.o., Brno
  - Fakultni Nemocnice Brno, Brno-Bohunice
  - Psychiatricka ambulance, Havířov
  - Psychiatricka Iecebna U Honzicka, Písek
  - Clintrial s.r.o., Prague
  - Psychiatricka Ambulance, Prague
  - Psychiaricka ambulance, Prague
  - Psychiatricka ambulance Prosek, Prague
  - Psychiatricke Centrum Praha, Prague 8-Bohunice
  - Psychosocialni Centrum, Přerov
  - Psychiatricka ambulance, Ústí nad Labem
- France (4):
  - CHS La Chartreuse-Pole 6, Dijon
  - Centre Hospitalier Specialise du Jura-Centre Medico Psychiatrique, Dole
  - Hopital Lapeyronie, Montpellier
  - CHRU de Nimes, Service de Psychiatrie adulte, Nîmes
- Hungary (7):
  - Obudai Egeszsegugyi Centurm Kft., Budapest
  - Fovarosi Onkormanyzat Szent Istvan Korhaz es Szent Laszlo Korhaz, Budapest
  - Kutvolgyi Klinikai Tomb SOTE IIIsz Belgyogyaszati Klinika, Budapest
  - Nyiro Gyula Korhaz, Budapest
  - Fovarosi Onkormanyzat Nyiro Gyula Korhaz, I. Pszichiatria, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaz, Gyula
- Japan (13):
  - Haruna Hospital, Shibukawa, Gunma
  - Goryokai Medical Corporation, Sapporo, Hokkaido
  - Sapporokousetsu Hospital, Sapporo, Hokkaido
  - Nagano Prefectural Mental Wellness Center-Komagane, Komagane, Nagano
  - Shonan Hospital, Matsumoto-shi, Nagano
  - Asakayama General Hospital, Sakai, Osaka
  - National Hospital Organization Hizen Psychiatric Center, Kanzaki, Saga-ken
  - Nishigahara Hospital, Kita-ku, Tokyo
  - Okehazama Hospital Fujita Kokoro Care Center, Aichi
  - Ongata Hospital, Hachioji, Tokyo
  - Yuge Hospital, Kumamoto
  - Arakaki Hospital, Okinawa
  - Kawada Hospital, Toyama
- Poland (5):
  - NZOZ Syntonia, Gdynia
  - NZOZ BioMed, Kielce
  - Wojewodzki Osrodek Lexznictwa Psychiatrycznego w Toruniu, Torun
  - Prywatny Gabinet Lekarski Jaroslaw Strzelec, Tuszyn
  - Przychodnia Lekarsko-Psychologiczna "Persona" Spolka Partnerska Lekarzy, Wroclaw
- Russia (6):
  - State Healthcare and Forensic Psychiatric Expertise Institution, Izhevsk
  - Nizhny Novgorod Regional State Institution of Healthcare, Nizhny Novgorod
  - St. Petersburg State Healthcare Institution (SPSHI), Saint Petersburg
  - St.Petersburg State Healthcare Institution (SPSHI), Saint Petersburg
  - St Petersburg State Government Healthcare Institution, Saint Petersburg
  - Mental Health Research Institute of Rams, Tomsk
- Serbia (5):
  - Clinical Centre of Serbia, Belgrade
  - Clinical Hospital Centre Dragisa Misovic, Belgrade
  - Psychiatric Clinic Clinical Center Kragujevac, Kragujevac
  - Clinical Centre Nis, Niš
  - Specialized Hospital for Psychiatric Diseased "Sveti Vracevi", Novi Kneževac
- Slovakia (2):
  - Vseobecna Nemocnica Rimavska Sobota, NaP, n.o. Bratislava, Rimavská Sobota
  - Psychiatricka ambulancia, Zlaté Moravce

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 2 phases in this study. In Phase 1 (Open-label Stabilization Phase), there was 1 reporting group. In phase 2 (Double-blind Maintenance Phase), there were 2 reporting groups.
  7 subjects completed the open-label but were not randomized DB(3- mood episode,3-not meeting the criteria for the DB phase,and 1-insufficient clinical response)
Groups:
- All Subjects: During the Open-label stabilization phase, subjects received flexible does of lurasidone 20 - 80 mg daily.
Period: Open Label Phase
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo | All Subjects
Started | 0 | 0 | 965
Completed | 0 | 0 | 503
Not Completed | 0 | 0 | 462
Not completed — Adverse Event | 0 | 0 | 59
Not completed — Lack of Efficacy | 0 | 0 | 107
Not completed — Lost to Follow-up | 0 | 0 | 76
Not completed — Protocol Violation | 0 | 0 | 45
Not completed — Withdrawal by Subject | 0 | 0 | 112
Not completed — Did not meet criteria for DB phase | 0 | 0 | 16
Not completed — Terminated at study completion | 0 | 0 | 5
Not completed — Mood episode | 0 | 0 | 42
Period: Double-Blind Phase
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo | All Subjects
Started | 246 | 250 | 0
Completed | 166 | 150 | 0
Not Completed | 80 | 100 | 0
Not completed — Adverse Event | 8 | 5 | 0
Not completed — Lost to Follow-up | 5 | 7 | 0
Not completed — Protocol Violation | 1 | 11 | 0
Not completed — Protocol Violation | 16 | 12 | 0
Not completed — Terminated at study completion | 2 | 0 | 0
Not completed — Recurrence of mood event | 48 | 64 | 0
Not completed — Administrative | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo | Total
Number analyzed (Participants) | 246 | 250 | 496
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 232 | 242 | 474
  >=65 years | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.43) | 43.2 (12.18) | 44.4 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 143 | 279
  Male | 110 | 107 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 38 | 79
  Not Hispanic or Latino | 205 | 212 | 417
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 21 | 44
  White | 213 | 216 | 429
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Argentina | 19 | 19 | 38
  Russian Federation | 30 | 31 | 61
  Hungary | 13 | 15 | 28
  United States | 73 | 76 | 149
  Japan | 5 | 5 | 10
  Czech Republic | 23 | 24 | 47
  Poland | 22 | 21 | 43
  Slovakia | 4 | 3 | 7
  Bulgaria | 20 | 20 | 40
  Chile | 9 | 11 | 20
  France | 8 | 6 | 14
  Serbia | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence of Mood Event During the Double Blind Treatment Phase
Description: A mood event is defined as one of the following during the double-blind phase:
  (1) Fulfilled Diagnostic and Statistical Manual of Mental Disorders, 4th Ed., Text Revision (DSM-IV-TR) criteria for manic, mixed manic, hypomanic, or depressive episode. (2) Required treatment intervention for manic, mixed manic, hypomanic, or depressive symptoms with any antipsychotic (other than study drug), antidepressant, mood stabilizer (other than lithium or divalproex), anxiolytic agents, benzodiazepine (beyond dosage allowed for anxiety, agitation, or insomnia). (3) Psychiatric hospitalization for any bipolar mood episode. (4) Young Mania Rating Scale (YMRS) or Montgomery-Asberg Depression Rating Scale (MADRS) total score ≥ 18 or Clinical Global Impression Bipolar Version, Severity of Illness (CGI BP S) score ≥ 4 at 2 consecutive assessments no more than 10 days apart. (5) Discontinuation from the study because of a mood event (as determined by the Investigator).
Time Frame: 28 weeks (up to 33 weeks)
Population: ITT (Intent to treat) population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 246 | 250
Days | NA [NA to NA] — not estimable due to an insufficient number of events | 207 [207 to NA] — not estimable due to an insufficient number of events
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; It was assumed that the recurrence event rates during the double-blind phase were to be 24% and 39% for subjects treated with lurasidone and placebo, respectively. A total of 120 recurrence events were required to achieve 90% power to detect the 15% difference in subjects who had a recurrence event during the double-blind phase between the treatment groups using a log-rank test with two sided alpha level of 0.05; Test type: Superiority or Other; p < 0.078, Cox Proportional Hazards Model — A hazard ratio of time to recurrence and its corresponding 95% Wald CI were estimated for the lurasidone arm vs.placebo arm, using a Cox proportional hazards model.Cox model included treatment effect as fixed effect, and stratified by pooled country; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.49 to 1.04]

2. Secondary Outcome: Time to All-cause Discontinuation
Time Frame: 28 weeks (up to 33 weeks)
Population: ITT population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 246 | 250
Days | 225 [204 to 233] | 207 [207 to 216]
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p < 0.034, Cox Proportional Hazards Model — A HR of time to discontinuation and corresponding 95% Wald CI were est. for lurasidone arm vs.the placebo arm, using a Cox proportional hazards model. Model included treatment effect including treatment as a fixed effect,stratified by pooled country; Cox Proportional Hazard = 0.72, 95% CI 2-sided [0.54 to 0.98]

3. Secondary Outcome: Time to Recurrence of a Manic, Mixed Manic, Hypomanic, or Depressed Episode
Time Frame: 28 weeks (up to 33 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 246 | 250
Days | NA [NA to NA] — not estimable due to an insufficient number of events | NA [207 to NA] — not estimable due to an insufficient number of events
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.113, Cox Proportional hazard Model — A HR of time to recurrence and its corresponding 95% Wald CI were estimated for lurasidone arm vs. placebo arm,using a Cox proportional hazards model. Model included treatment effect including treatment as a fixed effect stratified by pooled country; Cox Proportional Hazard = 0.72, 95% CI 2-sided [0.48 to 1.08]

4. Secondary Outcome: Percentage of Subjects Who Experience a Recurrence of a Manic, Mixed Manic, Hypomanic, or Depressed Episode
Time Frame: 28 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 246 | 250
percentage of participants | 16.7 | 21.6

5. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOCF) in CGI-BP-S Overall Score
Description: The CGI-BP-S overall score is a single value, clinician-rated assessment of overall bipolar illness severity and ranges from 1=Normal, not at all ill, to 7=Among the most extremely ill patients. a higher score is associated with greater illness severity.
Time Frame: Double-blind Baseline to week 28
Population: ITT population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. 2 lurasidone + Li/VPA subjects did not have post-DB baseline CGI-BP-S overall score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 244 | 250
units on a scale | 0.40 (0.085) | 0.49 (0.085)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.406, ANCOVA — analysis of ANCOVA model contains treatment ,pooled country, and mood stabilizer (lithium or divalproex) as fixed factors and baseline as a covariate; LS mean difference lurasidone vs.Placebo = -0.09, 95% CI 2-sided [-0.29 to 0.12]

6. Secondary Outcome: Change From Double -Blind Baseline to Week 28 (LOCF) in CGI-BP-S Mania Score
Description: The CGI-BP-S mania score is a single value, clinician-rated assessment of mania illness severity and ranges from 1=Normal, not at all ill to 7=Among the most extremely ill patients. A high score is associated with greater illness severity
Time Frame: Double-blind Baseline to week 28
Population: ITT population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. . 2 lurasidone + Li/VPA subjects did not have post-DB baseline CGI-BP-S mania score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 244 | 250
units on a scale | 0.10 (0.062) | 0.21 (0.062)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.162, ANCOVA — Analysis of Covariance (ANCOVA) model contains treatment, and pooled country, and mood stabilizer (lithium or divalproex) as fixed factors and baseline as a covariate; LS mean difference lurasidone vs.Placebo = -0.11, 95% CI 2-sided [-0.26 to 0.04]

7. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOCF) in CGI+-BP-S Depression Score
Description: The CGI-BP-S depression score is a single value, clinician-rated assessment of depression illness severity and ranges from 1=Normal, not at all ill to 7=Among the most extremely ill patients. A higher score is associated with a greater illness severity.
Time Frame: Double-blind Baseline to week 28
Population: ITT population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. 2 lurasidone + Li/VPA subjects did not have post-DB baseline CGI-BP-S depression score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 244 | 250
units on a scale | 0.35 (0.082) | 0.42 (0.081)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.496, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference lurasidone vs.Placebo = -0.07, 95% CI 2-sided [-0.27 to 0.13]

8. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOCF) in YMRS Total Score
Description: the YMRS is an 11-item instrument used to assess the severity of mania in subjects with a diagnosis of bipolar disorder. Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score). The YMRS total score is calculated as the sum of the 11 items. The YMRS total score ranges from 0 to 60. Higher scores are associated with greater severity of maia.
Time Frame: Double-blind Baseline to week 28
Population: ITT population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. . 2 lurasidone + Li/VPA subjects did not have post-DB baseline YMRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 244 | 250
units on a scale | 1.0 (0.43) | 1.8 (0.43)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.128, ANCOVA — Analysis of Covariance (ANCOVA) model contains treatment, and pool country, and mood stabilizer (lithium or divalproex) as fixed factors and baseline as a covariate; LS mean difference = -0.8, 95% CI 2-sided [-1.8 to 0.2]

9. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOCF) in MADRS Total Score
Description: The MADRS consists of 10 items, each rated on a Likert scale, from 0=Normal to 6=Most Severe. The MADRS total score is calculated as the sum of the 10 items. The MADRS total score ranges from 0 to 60. Higher scores are associated with greater severity of depressive symptoms.
Time Frame: Double-blind Baseline to week 28
Population: ITT population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. 2 lurasidone + Li/VPA subjects did not have post-DB baseline MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 244 | 250
units on a scale | 3.0 (0.57) | 3.5 (0.57)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.485, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference lurasdione vs.Placebo = -0.5, 95% CI 2-sided [-1.9 to 0.9]

10. Secondary Outcome: Change Fro Double-blind Baseline to Week 28 (LOCF) in QIDS-SR(16) Total Score
Description: The QIDS-SR16 is a 16-item self-report measure of depressive symptomatology which uses a computerized assessment interface for administration. The scoring system for the QIDS-SR16 converts responses to 16 separate items into nine DSM-IV symptom criterion domains. The nine domains comprise: depressed mood (Item 5); concentration/decision making (Item 10); self outlook (Item 11); suicidal ideation (Item 12); decreased interest (Item 13); decreased energy (Item 14); sleep disturbance (initial, middle, and late insomnia or hypersomnia) (highest score of Items 1 to 4); appetite/weight disturbance (highest score of Items 6 to 9); and psychomotor disturbance (highest score of Items 15 and 16). The QIDS-SR16 total score is calculated as the sum of the 9 domain scores. The QIDS-SR16 total score ranges from 0 to 27 with a high score indicating more severe symptoms.
Time Frame: Double-blind Baseline to week 28
Population: ITT population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. 7 lurasidone + Li/VPA subjects and 7 placebo +Li/VPA subjects did not have post-DB baseline QIDS-SR16 total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 239 | 243
units on a scale | 0.9 (0.27) | 1.1 (0.27)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.582, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference = -0.2, 95% CI 2-sided [-0.8 to 0.5]

11. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOF) in PANSS Positive Symptom (PANNS-P) Subscale Score
Description: The PANSS-P is a subset of items in the PANSS, an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS-P subscale score is the sum of the 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: Double-blind Baseline to week 28
Population: ITT Population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. . 6 lurasidone + Li/VPA subjects and 3 placebo +Li/VPA subjects did not have post-DB baseline PANSS-P score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 240 | 247
units on a scale | 0.2 (0.13) | 0.3 (0.13)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose; Test type: Superiority or Other; p = 0.420, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference lurasidone vs.Placebo = -0.01, 95% CI 2-sided [-0.5 to 0.2]

12. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOCF) in SDS Total Score
Description: The SDS is a composite of three self-rated items designed to measure the extent to which three major sectors in the patient's life are impaired by depressive symptoms. The SDS total score is calculated as the sum of the 3 items. The SDS total score ranges from 0 to 30. Higher scores are associated with greater severity of global functional impairments. If a subject has not worked/studied at all during the past week for reasons unrelated to the disorder, the SDS total score will be set to missing.
Time Frame: Double-blind Baseline to week 28
Population: ITT Population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on treatment they were randomized. 63 lurasidone + Li/VPA subjects and 57 placebo +Li/VPA subjects did not have post-DB baseline SDS total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 183 | 193
units on a scale | 0.4 (0.59) | 0.6 (0.61)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.788, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference lurasidone vs.Placebo = -0.2, 95% CI 2-sided [-1.6 to 1.2]

13. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOCF) in PIRS-2 Total Score
Description: The PIRS-2 is a 2-item self-report of insomnia assessed via a computer interface. Each item is scored from 0-3. The PIRS-2 total score is calculated as the sum of the 2 items. The PIRS total score ranges from 0 to 6. Higher scores are associated with greater severity of insomnia.
Time Frame: Double-blind Baseline to week 28
Population: ITT Population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. . 7 lurasidone + Li/VPA subjects and 7 placebo +Li/VPA subjects did not have post-DB baseline PIRS-2 total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 239 | 243
units on a scale | 0.4 (0.10) | 0.5 (0.10)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.380, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference lurasidone vs.Placebo = -0.1, 95% CI 2-sided [-0.3 to 0.1]

14. Secondary Outcome: Change From Double-blind Baseline to Week 28 (LOCF) in Q-LES-Q-SF Percent Maximum Possible Score
Description: The Q-LES-Q-SF is a 16-item self-report measure of the degree of enjoyment and satisfaction in various areas of daily living. The questionnaire was developed and validated for use in depressed outpatient subjects and has eight summary scales that reflect major areas of functioning: physical health, mood, leisure time activities, social relationships, general activities, work, household duties and school/coursework. Each item is rated on a 5-point scale, ranging from 1 (very poor) to 5 (very good). The Q-LES-Q-SF percentage maximum possible score is calculated as 100 × (Raw Score - 14 [Minimum Score]) / (70 [Maximum Score] - 14 [Minimum Score]). Higher percent maximum scores indicate better quality of life.
Time Frame: Double-blind Baseline to week 28
Population: ITT Population: all subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized. . 12 lurasidone + Li/VPA subjects and 11 placebo +Li/VPA subjects did not have post-DB baseline Q-LES-Q-SF percent maximum possible score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo
Number analyzed (Participants) | 234 | 239
units on a scale | -1.70 (1.022) | -2.07 (1.035)
Statistical Analysis 1: Comparison: Lurasidone 20-80 mg Flexible Dose vs Placebo; Test type: Superiority or Other; p = 0.772, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS mean difference lurasidone vs.Placebo = 0.37, 95% CI 2-sided [-2.14 to 2.88]

ADVERSE EVENTS:
Time Frame: For all subjects column: during open label phase (up to 20 weeks) For 7 lurasidone + Li/VPA and placebo +Li/VPA columns: during double blind phase (up to 28 weeks).
Description: During the open label phase there were 965 subjects There were three subjects that never received study drug and therefore are not included in this section
Groups:
- All Subjects: During the open-label stabilization phase, subjects received flexible does of lurasidone 20-80 mg daily
Arm/Group | Lurasidone 20-80 mg Flexible Dose | Placebo | All Subjects
Serious Adverse Events (participants affected / at risk) | 13/246 | 11/250 | 41/962
Other Adverse Events (participants affected / at risk) | 81/246 | 81/250 | 474/962
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20-80 mg Flexible Dose (N=246) | Placebo (N=250) | All Subjects (N=962)
Artiral fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Adominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecytitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 10 (10)
Mania (Psychiatric disorders) | 2 (2) | 3 (3) | 5 (5)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Bipolar 1 Disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Bipolar Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Intentional Self Injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Depressive Symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Acute Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Somatoform Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral edema (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) — Cerebral edema, 15 days, post - last dose, not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20-80 mg Flexible Dose (N=246) | Placebo (N=250) | All Subjects (N=962)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 111 (126)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 59 (66)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 53 (56)
Fatigue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 29 (30)
Nasopharyngitis (Infections and infestations) | 15 (17) | 12 (12) | 39 (45)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 9 (9) | 0 (0)
Weight Increased (Investigations) | 24 (24) | 13 (15) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 30 (30)
Headache (Nervous system disorders) | 21 (25) | 17 (21) | 88 (114)
Tremor (Nervous system disorders) | 15 (16) | 11 (12) | 43 (48)
Somnolence (Nervous system disorders) | 0 (0) | 4 (4) | 69 (75)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 34 (44)
Insomnia (Psychiatric disorders) | 9 (10) | 16 (25) | 77 (108)
Anxiety (Psychiatric disorders) | 4 (7) | 11 (17) | 41 (54)
Akathisia (Nervous system disorders) | 9 (10) | 8 (12) | 80 (91)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.